CLINICAL TRIAL: NCT06196411
Title: Effects of Task Oriented Training on Cognitive and Motor Functions in Patients With Stroke
Brief Title: Effects of Task Oriented Training in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HelinA
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Stroke; Task-oriented training; Bobath training; Motor functions; Cognitive functions
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Task-oriented Training Bobath Training
  Interventions: Behavioral: Task-oriented Training; Behavioral: Bobath Training
- Control Group (Active Comparator): Bobath Training
  Interventions: Behavioral: Bobath Training

INTERVENTIONS:
Behavioral: Task-oriented Training — Task-oriented training will be applied to study group 5 days a week, for a total of 6 weeks, in addition to Bobath training. Task-oriented training will consist of performing the lying, sitting, standing and walking exercises by performing tasks for specific goals. Exercises will be perform by accomplishing tasks such as touching the ball with the upper or lower extremities, reaching for the ball, crossing various tracks to move blocks from one place to another, walking through obstacles or climbing stairs.
  Arms: Study Group
Behavioral: Bobath Training — Bobath Concept includes sensory, perceptual and adaptive exercises aimed at improving function through mobilisation, weight-bearing, practicing more normal movement patterns and performing more efficient, less effortful tasks.

SUMMARY:
The aim of the randomized controlled study is to investigate the effects of task-oriented training on motor and cognitive functions combined with Bobath training in patients with stroke.

DETAILED DESCRIPTION:
Patients who meet the criteria will be informed about the study and volunteers will be included. When initial assessments will be completed, patients will be assigned to one of two possible sequences by simple randomization: study group (SG) or control group (CG).

All volunteers will recieve Bobath training program with the duration of 8 weeks. Additionally, task oriented training will be applied in SG, 5 days a week for 8 weeks.

All patients will be assessed in terms of motor functions and orientation, awareness, spatial perception, visuomotor construction, visual perception, praxis and thinking operations domains of cognitive funtions at the baseline and at the end of the study. Data will be collected from all the patients at baseline and at the end of the study (8 weeks) by the same physiotherapist who also will supervise the exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study
2. Be in the age range of 18-80 years
3. Clinical diagnosis of hemiplegia following stroke
4. Time since stroke between 2 and 8 weeks
5. Having stable vital signs
6. A score between 18-23 on the Mini Mental State Examination (MMSE)

Exclusion Criteria:

1. Having global aphasia and/or severe apraxia
2. Diagnosis of dementia or Alzheimer's prior to stroke
3. Participants who discontinued treatment
4. Receiving rehabilitation service before

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-24 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | 8 weeks
  The Mini Mental State Examination will be used for evaluating cognitive functions.
Dynamic Loewenstein Occupational Therapy Cognitive Assessment- Geriatric Version (DLOTCA-G) | 8 weeks
  DLOTCA-G is a battery test with a test booklet and test kits including 28 items in seven cognitive domains which are orientation, awareness, spatial perception, visuomotor construction, visual perception, praxis and thinking operations.
Functional Independence Measure (FIM) | 8 weeks
  FIM will be used to assess and rate motor and cognitive functional status in patients with stroke.
Barthel Index (BI) | 8 weeks
  BI will be used to assess motor functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Eksen Sağlık Inpatient Physical Therapy and Rehabilitation Center, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided